CLINICAL TRIAL: NCT05073367
Title: A Retrospective Observational Real-world Study to Evaluate Diagnosis Pattern, Treatment Pattern and Effectiveness of Eradication Treatment in Helicobacter Pylori (H. Pylori) Patients in China
Brief Title: A Study Reviewing Medical Records of Adults With Helicobacter Pylori Infections in China
Status: Completed | Type: Observational
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Other Study IDs: Vonoprazan-4008
Record Dates: First submitted 2021-10-08; First posted 2021-10-11 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Helicobacter Pylori
Keywords: Drug Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants with H. Pylori: Participants having evidence of H. pylori infection or having a positive result of H. pylori diagnostic testing recorded at inpatient or outpatient visits using pre-existing electronic medical record data in China will be observed retrospectively for 54 months.

SUMMARY:
The main aim of the study is to review treatment therapies in people with Helicobacter pylori (H. pylori) infections in standard hospital settings in China.

In this study, the study doctors will review medical records of participants who have had H. pylori infections any time from 1st January 2019 to 31st December 2021. This study is about collecting existing data only; participants are not treated and do not need to visit a study doctor during this study.

DETAILED DESCRIPTION:
This is a non-interventional, retrospective cohort study of participants who have evidence of H. pylori infection using pre-existing electronic medical record data in China. This study will evaluate the distribution of methods of eradication therapy among participants who received medications that were used in the eradication therapy for H. pylori infection.

Retrospective de-identified participant-level data will be collected primarily from hospitals in China between 1st January 2019 to 31st December 2021. The extracted electronic medical record dataset will include patient demographic information, visit information, diagnosis information, treatment information, and cost information (if available). All the participants will be assigned to a single observational cohort:

• Participants with H. pylori

This multi-center study will be conducted in China. The overall study duration will be approximately 54 months.

ELIGIBILITY:
Inclusion Criteria:

1. Participants with a record of H. pylori infection diagnosis or positive result of H. pylori diagnostic testing between 1st January 2019 and 31st December 2021.

Exclusion Criteria:

Not applicable.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult participants diagnosed with H. pylori infection or with positive record of H. pylori diagnostic testing will be included in this study.
Sampling Method: Probability Sample
Enrollment: 23000 (Actual)
Dates: Start 2022-09-21 (Actual); Primary Completion 2023-04-12 (Actual); Study Completion 2023-04-12 (Actual)

PRIMARY OUTCOMES:
Percentage of Each Eradication Regimen Initially Prescribed After Index Date | Up to 36 months
  Eradication therapy in this study includes standard bismuth quadruple therapy, standard triple therapy, and dual therapy. Eradication therapy will be identified according to the combination of drugs that are prescribed on the same day. Index date will be defined as first diagnosis date or the first date of a positive result of H. pylori diagnostic testing whichever came first during the participant identification period. For the percentage calculation of each eradication regimen, the denominator is the total usage count of all standard eradication therapies taken by eligible participants and the numerator is the total usage count of each eradication therapy.

SECONDARY OUTCOMES:
Percentage of Each Eradication Therapy's Treatment Duration From the Date of Prescription Until the Termination | From date of prescription up to 14 days
  Duration of eradication therapy is defined as the days in a medication-taking interval, which is equal to dosage by unit. Eradication therapy in this study includes standard bismuth quadruple therapy, standard triple therapy, and dual therapy. The duration of eradication therapy will be categorized into categorical variables including 7 days, 10 days, 14 days, or others. For percentage calculation of treatment duration of each eradication therapy, the denominator is the total usage count of all eradication therapies taken by eligible participants and the numerator is the count of the categorized duration of each eradication therapy.
Percentage of Each Diagnostic Testing Used Before the Prescription of Eradication Therapy | Up to 36 months
  H. pylori diagnostic testing includes non-invasive testing (urea breath testing [UBT], fecal antigen testing, serological testing) and invasive testing (polymerase chain reaction [PCR], culture, rapid urease test [RUT] and histology). For percentage calculation of each diagnosis before eradication therapy, the denominator is the total count of diagnostic testing and the numerator is the count of each type of diagnostic testing.
Percentage of Each Efficacy Evaluation Testing After the Termination of Eradication Therapy | Up to 36 months
  Efficacy evaluation testing is defined as H. pylori testing performed during the 28 days of efficacy evaluation period after treatment completion and this testing may extend to the follow-up period until observation period ends. For percentage calculation of efficacy evaluation testing after eradication therapy, the denominator is the total count of efficacy evaluation testing and the numerator is the count of each type of efficacy evaluation testing.
Percentage of the Duration From the Termination of Eradication Therapy Until the Efficacy Evaluation Testing | Up to 36 months
  The duration is defined as the time period between the last day of taking medication of eradication therapy and the day receiving efficacy evaluation testing. The duration of eradication therapy will be categorized into categorical variables including less than or equal to (<=) 4 weeks or greater than (>) 4 weeks. For percentage calculation of efficacy evaluation testing after each eradication therapy, the denominator is the total count of efficacy evaluation testing and the numerator is the count of duration (<=4 weeks or >4 weeks) .

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (5):
- China (5):
  - Shandong Provincial Hospital Affiliated to Shandong First Medical University, Jinan, Shandong
  - Shanghai Tenth Peoples Hospital, Shanghai, Shanghai Municipality
  - Army Medical Center of PLA, Chongqing, Sichuan
  - Tianjin First Central Hospital, Tianjin, Tianjin Municipality
  - Zhejiang Provincial Peoples Hospital, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- [Derived] Xu C, Pan W, Zhao Y, Li P, Zhou F, Xie L, Xu H. Diagnosis, Treatment Patterns and Eradication Success for Helicobacter pylori Infections in China: A Retrospective Observational Real-World Study. JGH Open. 2025 Oct 10;9(10):e70232. doi: 10.1002/jgh3.70232. eCollection 2025 Oct. PMID 41079532
- See also: To obtain more information on the study, click here/on this link — https://clinicaltrials.takeda.com/study-detail/61650ae4eb0e19002afd68c2